CLINICAL TRIAL: NCT01614314
Title: Dressing of Tunneled Central Venous Catheter: Preceptorship's Presence or Use of Auto-instructional Guide
Brief Title: Dressing of Tunneled Central Venous Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Fernanda Titareli Merizio Martins Braga, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CVCdressing
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Nursing Students
Keywords: Preceptorship, simulation, nursing, catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auto-instructional guide (Active Comparator): The subjects performed the procedure on a manikin simulator, with the aid of an auto-instructional guide, lasting one hour.
  Interventions: Other: Auto-instructional guide
- Preceptorship (Experimental): The subjects performed the procedure on a manikin simulator, with the aid of a nurse preceptorship, lasting one hour.
  Interventions: Other: Preceptorship

INTERVENTIONS:
Other: Preceptorship — After attending a lecture and a video on the dressing of the tunneled central venous catheter, the subjects performed the procedure on a manikin simulator, with the aid of a nurse preceptorship, lasting one hour.
  Arms: Preceptorship
Other: Auto-instructional guide — After attending a lecture and a video on the dressing of the tunneled central venous catheter, the subjects performed the procedure on a manikin simulator, with the aid of an auto-instructional guide, lasting one hour.
  Arms: Auto-instructional guide

SUMMARY:
The purpose of this study was to compare the performance of nursing undergraduates in dressing of tunneled central venous access in the simulator, according to the aid of a preceptorship or an auto-instructional guide.

DETAILED DESCRIPTION:
The simulation facilitates the acquisition of knowledge, skills and decision-making required for clinical practice. Mentoring has been employed and valued as pedagogical process qualifier.

The hypothesis of this study was that students who trained with the assistance of a preceptorship had better practical performance when compared to students who used an auto-instructional guide.

ELIGIBILITY:
Inclusion Criteria:

* students regularly enrolled in the last year of the undergraduate nursing program of a public university

Exclusion Criteria:

* students who did not comply with any of the study's phases
* students who presented performance > 70% in the pretest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Practical performance in carrying out dressing procedure | 1 day, immediately after the training simulator
  The practical performance in carrying out dressing procedure of each student was analyzed according to a list of 28 steps of procedure, including the preparation of environment and material, antisepsis, curative application and recording (score: 0 to 35). The list of items used to analyze the steps of the catheter dressing procedure were face and content validated by five experts working in the oncology field.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda TM Braga, PhD, RN, Principal Investigator — University of Sao Paulo at College of Nursing
Locations (1):
- University of Sao Paulo at College of Nursing, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Marmol MT, Braga FT, Garbin LM, Moreli L, dos Santos CB, de Carvalho EC. Central catheter dressing in a simulator: the effects of tutor's assistance or self-learning tutorial. Rev Lat Am Enfermagem. 2012 Nov-Dec;20(6):1134-41. doi: 10.1590/s0104-11692012000600016. English, Portuguese, Spanish. PMID 23258727